CLINICAL TRIAL: NCT01676870
Title: Exercise in Prevention of Metabolic Syndrome
Acronym: EX-MET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: Helse Stavanger HF (Other Government); Technical University of Munich (Other); The University of Queensland (Other); KJ Fisiosport (Unknown); University of Sao Paulo (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2011/1230
Record Dates: First submitted 2012-08-29; First posted 2012-08-31 (Estimated); Last update posted 2020-02-07 (Actual); Status verified 2020-02

CONDITIONS: Metabolic Syndrome
Keywords: exercise training; exercise therapy; physical fitness; risk factors
MeSH Terms: conditions — Metabolic Syndrome

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1x4 aerobic interval training (Experimental): 1x4min aerobic interval training (1-AIT), 3 times a week
  Interventions: Behavioral: 1x4 aerobic interval training
- 4x4 aerobic interval training (Experimental): 4x4min aerobic interval training (4-AIT), vigorously exercise according to today's guidelines, 3 times a week
  Interventions: Behavioral: 4x4 aerobic interval training
- traditional moderate training (Active Comparator): traditional moderate training (CME), moderate exercise at least 30 min, 5 days a week or more, according to today's guidelines
  Interventions: Behavioral: traditional moderate training

INTERVENTIONS:
Behavioral: 1x4 aerobic interval training — endurance training as walking/running "uphill" 3 times/week for 16 weeks (2 supervised sessions (treadmill) and 1 at home each week) at 90% of Hfmax. Warm-up 10 min at 70% of maximal heart frequency (Hfmax), 5min cool-down.
  Arms: 1x4 aerobic interval training
Behavioral: 4x4 aerobic interval training — endurance training as walking/running "uphill" 3 times/week for 16 weeks (2 supervised sessions (treadmill) and 1 at home each week) at 90% of Hfmax. Warm-up 10 min at 70% of maximal heart frequency (Hfmax), 3 min active pause between each interval, 5min cool-down.
  Arms: 4x4 aerobic interval training
Behavioral: traditional moderate training — moderate intensity treadmill training (50-70% of HRmax) for a minimum of 30min, 5 times a week for 16 weeks (2 supervised sessions and 3 or more home).
  Arms: traditional moderate training

SUMMARY:
The primary objective of the study is to compare in a real-world setting the efficacy of traditional training (today's guideline, vigorously or moderate exercise) and amount of aerobic interval training (1-AIT) in reduction of risk factors constituting metabolic syndrome.

The secondary objective is to compare the efficacy of traditional moderate training (today's guideline) and amount of aerobic interval training (1-AIT vs. 4-AIT) in improving aerobic capacity, cardiovascular function, skeletal muscle contractile function, skeletal muscle energy metabolism, left ventricle systolic and diastolic function at rest and right ventricular function.

The investigators hypothesized that aerobic interval training would reverse features of the metabolic syndrome more than traditional training.

DETAILED DESCRIPTION:
This study describes a randomized multicenter clinical trial designed to test the hypothesis that a 16-week program, with one year follow up of vigorously exercise defined from today's guidelines (performed as 4-AIT (4x4min aerobe interval training)) yields larger beneficial effects in reducing risk factors constituting the metabolic syndrome than continuously moderate intensity exercise (CME) defined from today's guidelines.

Furthermore, the importance of the amount of aerobic interval training remains unclear and it is unknown how little "one can get away with" and still obtain substantial beneficial cardiovascular effects. Therefore, the investigators will also determine whether one bout of aerobe interval training (AIT) - 1-AIT = 1x4min aerobe interval training, can give beneficial effects compared to 4-AIT and CME.

Evaluation criteria are risk factors constituting metabolic syndrome, aerobic capacity measured as peak oxygen uptake and compliance to intervention. Assessments will be made before and after the 16-week program, and at six month, and 1 and 3 years follow-up. According to estimates based on data from previously studies, 3, 4 a total number of 465 patients randomized 1:1:1 to the three interventions gives 80% power to detect an effect of 4-AIT compared to 1-AIT/CME of 51% recovery versus 37% recovery from metabolic syndrome at the 5% significance level.

ELIGIBILITY:
Inclusion Criteria:

* metabolic syndrome defined according to the IDF-criteria

Exclusion Criteria:

* unstable angina
* recent cardiac infarction (4weeks)
* uncompensated heart failure
* severe valvular illness
* pulmonary disease
* uncontrolled hypertension
* kidney failure
* orthopedic/neurological limitations
* cardiomyopathy
* planned operations during the research period
* reluctant to sign the consent form
* drug or alcohol abuse
* participants in a parallel study

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Actual)
Dates: Start 2012-01 (Actual); Primary Completion 2019-12-15 (Actual); Study Completion 2019-12-15 (Actual)

PRIMARY OUTCOMES:
cardiovascular risk factors constituting metabolic syndrome | up to 3 years
  Endothelial function and blood pressure, biopsies from the m. vastus lateralis, Protein and expression levels, oxidized LDL and adiponectin in blood plasma

CONTACTS AND LOCATIONS:
Overall Officials: Ulrik Wisløff, PhD prof, Study Director — Norwegian University of Science and Technology
Locations (6):
- School of Human Movement Studies, University of Queensland, Saint Lucia, Australia
- University of Sao Paulo, São Paulo, Brazil
- KJ Fisioterapi, Guayaquil, Ecuador
- Internal Medicine, Cardiology, Sports Medicine Chair Dep. Prevention, Rehabilitation and Sports Medicine Faculty of Medicine University Hospital, Munich, Germany
- Norway (2):
  - Stavanger University Hospital, Stavanger
  - St. Olavs hospital, Trondheim

REFERENCES:
- [Background] Tjonna AE, Ramos JS, Pressler A, Halle M, Jungbluth K, Ermacora E, Salvesen O, Rodrigues J, Bueno CR Jr, Munk PS, Coombes J, Wisloff U. EX-MET study: exercise in prevention on of metabolic syndrome - a randomized multicenter trial: rational and design. BMC Public Health. 2018 Apr 2;18(1):437. doi: 10.1186/s12889-018-5343-7. PMID 29609582
- [Derived] Ramos JS, Dalleck LC, Fennell M, Martini A, Welmans T, Stennett R, Keating SE, Fassett RG, Coombes JS. Exercise Training Intensity and the Fitness-Fatness Index in Adults with Metabolic Syndrome: A Randomized Trial. Sports Med Open. 2021 Dec 24;7(1):100. doi: 10.1186/s40798-021-00395-7. PMID 34951682
- [Derived] Ramos JS, Dalleck LC, Borrani F, Beetham KS, Wallen MP, Mallard AR, Clark B, Gomersall S, Keating SE, Fassett RG, Coombes JS. Low-Volume High-Intensity Interval Training Is Sufficient to Ameliorate the Severity of Metabolic Syndrome. Metab Syndr Relat Disord. 2017 Sep;15(7):319-328. doi: 10.1089/met.2017.0042. Epub 2017 Jun 22. PMID 28846513
- [Derived] Ramos JS, Dalleck LC, Borrani F, Mallard AR, Clark B, Keating SE, Fassett RG, Coombes JS. The effect of different volumes of high-intensity interval training on proinsulin in participants with the metabolic syndrome: a randomised trial. Diabetologia. 2016 Nov;59(11):2308-2320. doi: 10.1007/s00125-016-4064-7. Epub 2016 Aug 1. PMID 27480182